CLINICAL TRIAL: NCT01461343
Title: Evaluation of Pulmonary Perfusion Heterogeneity and Compliance in Patients With Pulmonary Arterial Hypertension Using Functional Positron Emission Tomography Imaging
Brief Title: Evaluation of Pulmonary Perfusion Heterogeneity and Compliance in Patients With Pulmonary Hypertension Using Positron Emission Tomography Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert Scott Harris, M.D., Associate Physician, Massachusetts General Hospital; Assistant Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011-P-001880/1
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension, PET imaging, CT/PET
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pulmonary hypertension (Experimental): Patients with Group I pulmonary arterial hypertension and exercise-induced pulmonary hypertension to undergo CT imaging, functional PET imaging
  Interventions: Other: CT imaging, functional PET imaging
- healthy controls (Active Comparator): healthy adults to serve as controls and to undergo the same study procedures: CT imaging, functional PET imaging
  Interventions: Other: CT imaging, functional PET imaging

INTERVENTIONS:
Other: CT imaging, functional PET imaging — Physiology study using CT and functional PET imaging with 13NN and 11CO as radiotracers; images obtained before and after administration of inhaled nitric oxide and balance 80% oxygen as pulmonary vasodilators

SUMMARY:
The purpose of the study is to find out how the blood flow changes in the lungs of people with pulmonary hypertension compared to healthy individuals without pulmonary hypertension. We would like to find out if there are differences in how blood flows when subjects are given a drug to dilate (widen) the arteries in their lungs and when they breathe extra oxygen. We will compare the results to when subjects don't receive any drug or extra oxygen. We hope that knowing about these differences will help us to better understand pulmonary hypertension and how to diagnose it earlier.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) refers to abnormalities in the pulmonary vasculature associated with a diverse group of disorders. The World Health Organization (WHO) classifies pulmonary hypertension into five groups, with Group I comprising pulmonary arterial hypertension (formerly referred to as "primary pulmonary hypertension"). Although not currently a part of the WHO classification, exercise-induced pulmonary arterial hypertension (EIPAH), defined by normal pulmonary artery pressures at rest and elevation of pulmonary pressures with exercise, is increasingly recognized as a distinct clinical entity. In some patients, exercise-induced pulmonary hypertension may represent a precursor for developing an established elevation in pulmonary pressures at rest that defines PAH. Functional PET imaging has not previously been utilized to quantify perfusion and vascular compliance in patients with pulmonary arterial hypertension. The overall goal of this study is to evaluate regional lung perfusion, perfusion heterogeneity, and vascular compliance in patients with both exercise-induced and resting pulmonary hypertension using functional positron emission tomography imaging. Ultimately, if quantifiable differences between healthy subjects and patients with PAH are detected with 13NN and 11CO labeled PET, functional PET imaging may provide a useful imaging modality in early diagnosis of pulmonary hypertension and monitoring response to therapy. In this pilot study, we will recruit 10 adult patients with pulmonary hypertension (5 with PAH and 5 with EIPAH) who are on stable PAH-specific therapy (if any), and 5 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* General

  1. A signed and dated written informed consent is obtained from the subject.
  2. The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  3. Available to complete the study.
  4. Able to lie flat and able to perform a 30 second breath hold.
* Patients with Pulmonary Hypertension

  1. Subject is male or female aged = or > 18 years of age and < or = 70 years.
  2. Subject is diagnosed with pulmonary arterial hypertension (WHO Group I, by right heart catheterization, mean PA pressure > 25 and PCWP < 15) or exercise-induced pulmonary hypertension (by right heart catheterization + Level III cardiopulmonary exercise testing, mean PAP > 30 and PCWP < 20 during exercise, but normal at rest), with the most recent of above diagnostic tests taking place within 12 months of study entry.
  3. If patient has been on PAH-specific therapy, the therapy (agent and dose) has been unchanged for at least 3 months.

Exclusion Criteria:

* General

  1. FEV1 and/or TLC < 70% predicted
  2. PCWP > 15 mm Hg
  3. Inability to perform the study (by primary MD or investigator assessment)
  4. Subjects who have a past or present disease, which as judged by the Investigators may affect the outcome of this study
  5. The subject has suspected history of drugs or alcohol abuse within the six months prior to the screening visit.
  6. The subject has a positive pregnancy test.
  7. The subject is unable to perform the respiratory manoeuvres necessary for the exam.
  8. The subject has been exposed to a radiation dose over the past year that, when added to the radiation dose expected in this study, would exceed permissible yearly exposure as determined by the MGH radiation safety committee.
* Subjects with Pulmonary Hypertension

  1. Subject with clinical instability in the judgment of the investigator, or hospitalization for progression of pulmonary hypertension or right heart failure in the three months prior to the study.
  2. Subjects in whom PAH therapy has been escalated (additional agent started) within 3 months of enrolment.
  3. Subject with diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, allergic rhinitis, asthma, or COPD.
  4. Subject that had a respiratory tract infection in the 4 weeks prior to the screening visit and throughout the duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2017-11-21 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of perfusion | One imaging visit lasting up to 3 hours
  Images will be generated with positron emission tomography that will be used to calculate the degreee to which the blood flow in the lung is patchy rather than smooth. The statistical measure of this is called the coefficient of variation.

SECONDARY OUTCOMES:
Vascular compliance | One imaging visit lasting up to 3 hours
  Positron emission tomography images will be obtained during different phases of the heart beat that will show how the blood vessels in the lung stretch with ejection of blood from the heart. The change in volume of the blood vessels is called vascular compliance and is a measure of blood vessel stiffness.
Perfusion gradient | One imaging visit lasting up to 3 hours
  From the images of blood flow in the lung, the change in mean blood flow from the bottom of the lung to the top will be calculated. Normally, there is more blood flow at the bottom of the lung compared to the top, but this can be changed with lung disease.

CONTACTS AND LOCATIONS:
Overall Officials: R. Scott Harris, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States